CLINICAL TRIAL: NCT06781385
Title: Intra-Arterial Tenecteplase Following Endovascular Thrombectomy for Large Vessel Occlusion Stroke
Acronym: TNK-FLOW
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00121066; 40010317 (Other: Genentech, Inc)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke
Keywords: brain hemorrhage; stroke; blood clot
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages; Stroke; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-arterial Tenecteplase (Experimental): Following endovascular thrombectomy for large vessel occlusion stroke one-time dose of intra-arterial Tenecteplase (0.125 mg/kg, maximum dose 12.5 mg) will be delivered over 5-10 seconds by the treating neuro-interventionalist through a microcatheter positioned as close as possible to the residual thrombus or as distal as possible in the originating vessel, per the discretion of the neuro-interventionalist.
  Interventions: Drug: Intra-arterial Tenecteplase
- Intra-arterial Saline (Placebo Comparator): Following endovascular thrombectomy for large vessel occlusion stroke one-time dose of saline (0.9% NaCl solution) will be delivered over 5-10 seconds by the treating neuro-interventionalist through a microcatheter positioned as close as possible to the residual thrombus or as distal as possible in the originating vessel, per the discretion of the neuro-interventionalist.
  Interventions: Drug: Intra-arterial Saline

INTERVENTIONS:
Drug: Intra-arterial Tenecteplase — One-time dose of intra-arterial tenecteplase post-thrombectomy
  Arms: Intra-arterial Tenecteplase
Drug: Intra-arterial Saline — One-time dose of intra-arterial saline post-thrombectomy
  Arms: Intra-arterial Saline

SUMMARY:
The purpose of this study is to determine the safety and feasibility of using intra-arterial Tenecteplase in patients undergoing blood clot extraction for treatment of acute ischemic (non-bleeding) stroke. Intravenous Tenecteplase is FDA-approved to treat patients with an ischemic stroke presenting within the 0-3-hour time window.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the safety and feasibility of intra-arterial Tenecteplase in selected patients with persistent post-thrombectomy hypoperfusion on computed tomography perfusion based on symptomatic intracranial hemorrhage (parenchymal hematoma type 2, subarachnoid hemorrhage, and/or intraventricular hemorrhage producing decline from the initial NIHSS of ≥ 4 points) at 24-36 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient/legally authorized representative has signed the Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Functionally independent (modified Rankin scale 0-2) prior to presentation
* Baseline National Institutes of Health Stroke Scale (NIHSS) ≥ 6
* Clinical syndrome consistent with occlusion of the internal carotid artery (ICA) or proximal middle cerebral artery (MCA), presenting within 4.5- to 24-hours of TLKW
* Evidence of ICA, MCA-M1, or MCA-M2 occlusion on baseline computed tomography angiogram (CTA) or magnetic resonance angiogram (MRA). ICA/MCA tandem occlusions may be enrolled
* Alberta Stroke Program Early Computed Tomography Score ≥ 6 on pre-thrombectomy unenhanced CT as determined by treating neurologist or reading radiologist
* Pre-thrombectomy computed tomography perfusion (CTP) or magnetic resonance perfusion (MRP) with core infarction (cerebral blood flow < 30%) < 70 ml, mismatch ratio ≥ 1.8, mismatch volume ≥ 15 ml (completed within 120 minutes of skin puncture for thrombectomy)
* Endovascular thrombectomy of ICA, MCA-M1 or MCA-M2 occlusion performed according to local standard of care, defined as at least completing the initial diagnostic angiogram
* CTP performed with RAPID AI AngioFlowTM within 30 minutes of thrombectomy completion
* Modified thrombolysis in cerebral infarction (mTICI) 2b-3 revascularization following endovascular thrombectomy (EVT) (or after initial diagnostic angiogram)
* Presence of Tm > 6 lesion on post-EVT CTP of adequate quality for interpretation in the distribution of the symptomatic occlusion

Exclusion Criteria:

* Current participation in another investigational drug or device study
* Known hypersensitivity or allergy to any ingredients of tenecteplase
* Active internal bleeding
* Known bleeding diathesis (e.g., Alzheimer's patients taking lecanemab)
* Systolic blood pressure > 185 mm Hg or diastolic blood pressure > 110 mm Hg after EVT, refractory to medical therapy
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; recent oral anticoagulant therapy with INR > 1.7
* Use of one of the new oral anticoagulants within the last 48 hours (dabigatran, rivaroxaban, apixaban, edoxaban)
* Treatment with a thrombolytic within the last 3 months prior to randomization
* Baseline platelet count < 100,000/mcL (results must be available prior to treatment)
* Baseline blood glucose > 400 mg/dL (22.20 mmol/L)
* Baseline blood glucose < 50 mg/dL; needs to be normalized prior to randomization
* Intracranial or intraspinal surgery or trauma within 2 months
* Intracranial malignant neoplasm, arteriovenous malformation, or unsecured aneurysm > 1 cm
* Other serious, advanced, or terminal illness (investigator's judgment) or life expectancy is less than 6 months
* History of acute ischemic stroke in the last 90 days
* History of hemorrhagic stroke
* Presumed septic embolus; suspicion of bacterial endocarditis
* Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the patient if an endovascular procedure was to be performed
* Pregnant
* Acute intracranial hemorrhage on pre-thrombectomy imaging or suspected acute intracranial hemorrhage after EVT
* Acute bilateral strokes on initial imaging
* Multiple acute intracranial occlusions (except ICA/MCA) on initial CTA or MRA
* Significant hemispheric mass effect or any amount of midline shift due to acute stroke
* Placement of cervical carotid or intracranial stent during thrombectomy procedure requiring dual antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participants with Change in Symptomatic Intracranial Hemorrhage | Hour 36
  Number of participants with symptomatic intracranial hemorrhage (parenchymal hematoma type 2, subarachnoid hemorrhage, and/or intraventricular hemorrhage) producing decline from the initial National Institutes of Health Stroke Scale (NIHSS) of ≥ 4 points.
Participants with Parenchymal Hematoma Type 1 | 24 Hours
  Number of participants with parenchymal hematoma type 1
Participants with Parenchymal Hematoma Type 2 | 24 Hours
  Number of participants with parenchymal hematoma type 2
30-Day Mortality Count | Day 30
  Number of patients expired
90-Day Mortality Count | Day 90
  Number of patients expired
Number of Grade 3 Adverse Events | Hour 24
  Total number of grade 3 adverse events
Number of Grade 3 Adverse Events | Day 5
  Total number of grade 3 adverse events
Number of Grade 3 Adverse Events | Day 30
  Total number of grade 3 adverse events
Number of Grade 3 Adverse Events | Day 90
  Total number of grade 3 adverse events

OTHER OUTCOMES:
Proportion of subjects achieving early neurological improvement | Hour 24
  Proportion of subjects achieving early neurological improvement, defined as National Institutes of Health Stroke Scale (NIHSS) reduction by ≥ 4 points or total NIHSS 0-2
Proportion of subjects achieving delayed neurological improvement | Day 30, Day 90
  Proportion of subjects achieving delayed neurological improvement, defined as National Institutes of Health Stroke Scale (NIHSS) reduction by ≥ 4 points or total NIHSS 0-2
Ordinal Modified Rankin Scale score | Day 90
  Modified Rankin scale scores range from 0-6. Higher score indicates greater disability.
Participants with Change in Modified Rankin Scale Score 0-2 Points | Day 90
  Number of participants with change in Modified Rankin Scale score of 0-2 points or return to baseline modified Rankin scale score.
Participants with Change in Modified Rankin Scale Score 0-1 Points | Day 90
  Number of participants with change in Modified Rankin Scale score of 0-1 points or return to baseline modified Rankin scale score.
Participants with Change in Modified Rankin Scale Score 0-3 Points | Day 90
  Number of participants with change in Modified Rankin Scale score of 0-3 points or return to baseline modified Rankin scale score.
Change in Infarct Volume | Hour 24
  Change in infarct volume on follow up CT or MRI
Barthel Index Score | Day 90
  Number of participants with Barthel Index score ≥ 95.
Median EuroQol-5-Dimension (EQ-5D) Index | Day 90
  Median EuroQol-5-Dimension (EQ-5D) index has a score range of -0.573 to 1. Higher score indicates better quality score.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Karamchandani, MD, Principal Investigator — Atrium Health Neurosciences Institute
Locations (1):
- Atrium Health Neurosciences Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No